CLINICAL TRIAL: NCT06238960
Title: Effectiveness of Telerehabilitation in Continuity With Outpatient Physiotherapy After Total Hip Replacement: Randomized Clinical Trial.
Brief Title: Effectiveness of Telerehabilitation in Continuity With Outpatient Physiotherapy After Total Hip Replacement.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TELERIABPTA
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Total Hip Replacement; Telerehabilitation; Physiotherapy
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): the patients who will be randomized and subjected to the experimental treatment will undergo a physiotherapy treatment with a biweekly frequency which will be started at the same times as the standard group.
  After the sixth session, the process will continue through telerehabilitation until the end of outpatient treatment.
  Interventions: Other: Telerehabilitation
- traditional physiotherapy (Active Comparator): Patients who will be randomized and subjected to standard treatment (usual care at our clinic) will undergo physiotherapy treatment on a bi-weekly basis in person.
  Interventions: Other: Traditional rehabilitation

INTERVENTIONS:
Other: Telerehabilitation — the patient will undergo 10 session of tele rehabilitation in continuity with traditional physiotherapy
  Arms: Telerehabilitation
Other: Traditional rehabilitation — the patient will undergo 16 session of outpatient physiotherapy rehabilitation
  Arms: traditional physiotherapy

SUMMARY:
Total arthroplasty (THA) is the treatment of choice for severe osteoarthritis of the hip joint. Following this type of intervention, a multidisciplinary rehabilitation approach allows you to reduce pain and improve the ability to carry out activities of daily living (ADL), but it is not clear what the optimal rehabilitation program is. Recently, the use of telerehabilitation has increased over the years. Specifically, in treatment of patients following THA surgery, telerehabilitation is able to give similar results to the treatment performed in person terms of pain and function. The aim of this study is to verify whether telerehabilitation associated with In-person treatment is comparable in terms of pain, recovery functionality and patient participation and satisfaction, compared to those provided by rehabilitation alone in the presence of patients undergoing THA surgery.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone total hip replacement surgery (THA)
* Start outpatient treatment within 7 days of discharge from the Orthopedic Department
* Age between 50 and 80 years.
* Continuation of rehabilitation treatments at the IOR Physical Medicine and Rehabilitation service in Argenta.
* The subjects or any caregivers must be able to use an electronic device (PC, tablet, smartphone).

Exclusion Criteria:

* patients undergoing revision of previous prosthesis surgery
* difficulty understanding the Italian language/language barrier
* unavailability stable wi-fi connection by the patient

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-02-10 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Hip disability and Osteoarthritis Outcome score (HOOS) | At baseline (day 0)
  The HOOS is a 40-item self-report questionnaire with 5 subscales. A normalized score is calculated for each subscale with 0 indicating extreme symptoms and 100 representing no symptoms.
Hip disability and Osteoarthritis Outcome score (HOOS) | After 8 weeks
  The HOOS is a 40-item self-report questionnaire with 5 subscales. A normalized score is calculated for each subscale with 0 indicating extreme symptoms and 100 representing no symptoms.
Hip disability and Osteoarthritis Outcome score (HOOS) | After 12 weeks
  The HOOS is a 40-item self-report questionnaire with 5 subscales. A normalized score is calculated for each subscale with 0 indicating extreme symptoms and 100 representing no symptoms.

SECONDARY OUTCOMES:
Timed Up and GO (TUG) | After 8 weeks
  The test measures the time (in seconds) it takes a patient to get up from a chair, walk 3 meters, reverse and sit back in the chair. It can be performed without aids or with the aid usually used by the patient to walk.
Timed Up and GO (TUG) | After 12 weeks
  The test measures the time (in seconds) it takes a patient to get up from a chair, walk 3 meters, reverse and sit back in the chair. It can be performed without aids or with the aid usually used by the patient to walk.
Harris Hip Score (HHS) | After 8 weeks
  a multi-disability measurement tool, validated and translated into Italian, composed of a questionnaire and a specific clinical examination which has the aim of evaluating ADL and function in subjects with hip pathology
Harris Hip Score (HHS) | After 12 weeks
  a multi-disability measurement tool, validated and translated into Italian, composed of a questionnaire and a specific clinical examination which has the aim of evaluating ADL and function in subjects with hip pathology

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto ortopedico Rizzoli, Bologna, Italia, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Sadiq S, Ahmad A, Ahmed A, Khan I, Asim HM, Aziz A. Role of tele-rehabilitation in patients following total hip replacement: Systematic review of clinical trials. J Pak Med Assoc. 2022 Jan;72(1):101-107. doi: 10.47391/JPMA.832. PMID 35099447
- [Result] Nelson M, Bourke M, Crossley K, Russell T. Telerehabilitation is non-inferior to usual care following total hip replacement - a randomized controlled non-inferiority trial. Physiotherapy. 2020 Jun;107:19-27. doi: 10.1016/j.physio.2019.06.006. Epub 2019 Jun 25. PMID 32026820